CLINICAL TRIAL: NCT03476863
Title: IMPACT OF ALVEOLAR RECOVERY MANEUVER ON PULMONARY FUNCTION AND RESPIRATORY MECHANISM IN PATIENTS SUBMITTED TO BARIATRIC SURGERY ASSESSED BY ELECTROMAT IMPEDANCE TOMOGRAPHY: A RANDOMIZED CLINICAL TRIAL
Brief Title: Gastroplasty and Electrical Impedance Tomography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Daniella Cunha Brandao (Other)
Collaborators: Antonio Christian Evangelista Gonçalves (Unknown); Armèle Dornelas de Andrade (Unknown); Norma Sueli Pinheiro Módolo (Unknown)
Responsible Party: Sponsor-Investigator, Daniella Cunha Brandao, PhD, Universidade Federal de Pernambuco
Organization: Universidade Federal de Pernambuco (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Gastro01
Record Dates: First submitted 2018-03-09; First posted 2018-03-26 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Gastropathy
MeSH Terms: conditions — Stomach Diseases

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alveolar Recruitment Maneuver (Experimental)
  Interventions: Procedure: Alveolar Recruitment Maneuver
- Conventional mechanical ventilation (Active Comparator)
  Interventions: Procedure: Conventional mechanical ventilation

INTERVENTIONS:
Procedure: Alveolar Recruitment Maneuver — Patients in the Experimental Group will be submitted to ARM, immediately after abdominal desinflation of the pneumoperitoneum (PNP). The ARM will be performed with PEEP of 15 cmH2O for thirty seconds, 20 cmH2O for thirty seconds, 25 cmH2O for thirty seconds, 30 cmH2O for one minute and a inspiratory plateau pressure of 15 cmH2O above PEEP, totaling two minutes and thirty seconds.The data of the TIE will be continuously recorded and the hemodynamic and respiratory function variables such as heart rate (HR), respiratory rate (RF), mean arterial pressure (MAP), peripheral oxygen saturation (SpO2) and final gas expiratory pressure carbon dioxide (PETCO2) will be recorded in several moments: immediately after the monitoring, and the patient is still on spontaneous ventilation, 5min after orotracheal intubation, after the installation of the pneumoperitoneum, before and after the execution of the MRA and in the Post-OP, in the first 24h, along with new lung function tests.
  Arms: Alveolar Recruitment Maneuver
Procedure: Conventional mechanical ventilation — Immediately after intubation, patients will undergo mechanical ventilation with the ventilator (Dixtal DX 5020) in volume controlled mode with an ideal tidal volume of 7 ml / kg body weight, a set frequency to maintain a carbon dioxide of 35-42 mmHg, and an inspiratory / expiratory ratio of 1: 2. The inspiratory oxygen fraction (FIO2) will be 0.5.
  Arms: Conventional mechanical ventilation

SUMMARY:
Worldwide there is a high prevalence of morbid obesity with a progressive increase in incidence in recent years, causing serious consequences for the health services. Approximately 12% of the world population is obese and Brazil is in 77º without world ranking of countries in cases of obesity. In this context, bariatric surgery appears as an effective method of treating refractory obesity. Support of high fractions of oxygen administered during anesthesia is produced, it accepts the use of Positive Positive Positive Pressure (PEEP) through the Alveolar Recruitment Maneuver (ARM), which has been used allowing small fractions inspired by oxygen, which reduces intra-and postoperative atelectasis and optimizes gas exchange during anesthesia. In order to better monitor ventilatory mechanics, Electrical Impedance Tomography (EIT) appears as a cheap imaging method when compared to a non-invasive magnetic resonance imaging (CT) or MRI, with no side effects and recent studies shown in its life as pneumothorax , MRA monitoring, collapse detection, and PEEP titration. The aim of this study is to evaluate the impact of ARM and its repercussions on lung function and respiratory mechanics. This is a randomized controlled clinical trial with patients undergoing videolaparoscopic gastroplasty surgery, of both sexes. Patients were randomly assigned to Control Group and Experimental Group. Patient evaluation is performed without before, during and postoperative, through a pulmonary function test and EIT.

ELIGIBILITY:
Inclusion Criteria:

* Patients submitted to videolaparoscopy gastroplasty surgery, of both sexes

Exclusion Criteria:

* Severe pneumopathies;
* Congestive heart failure (NYHA class III or IV);
* Coronary artery disease, and those who, for any clinical, surgical and psychosocial reasons, require intervention by laparotomy and those with hemodynamic instability (PAM) <60 mmHg) at the time recorded for performing the alveolar recruitment maneuver.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2018-03-23 (Actual); Primary Completion 2018-03-25 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Pulmonary aeration by electrical impedance tomography | 2 days
  The TIE will evaluate the behavior of regional pulmonary aeration by measuring the electrical impedance variation throught the mean electrical impedance at the end of expiration (MIEFE) and the mean electric impedance at the end of the (MIEFI). Thirty-two electrodes will be attached circumferentially (equally spaced) around the volunteer's chest, just below the level of the axilla. An electric current of 5 mA will be emitted at 125 KHz by means of a pair of electrodes.
  The data evaluated by the TIE will be recorded before, during and immediately after performing the maneuvers until the reduction to the baseline values is verified.
regional pulmonary ventilation by measuring the electrical impedance variation | 2 days
  The TIE will evaluate the behavior of regional pulmonary ventilation by measuring the electrical impedance variation (ΔZ = inspiratory impedance - expiratory impedance) of the distribution of regional pulmonary ventilation in the dependent and nondependent regions of the right and left lungs, and the dynamic compliance of the respiratory system.
  Thirty-two electrodes will be attached circumferentially (equally spaced) around the volunteer's chest, just below the level of the axilla. An electric current of 5 mA will be emitted at 125 KHz by means of a pair of electrodes.
  The data evaluated by the TIE will be recorded before, during and immediately after performing the maneuvers until the reduction to the baseline values is verified.

SECONDARY OUTCOMES:
Pulmonary Function | 2 days
  To measure the spirometric values, 3 maneuvers will be performed according to American Thoracic Society Guidelines recommendations, with the participant sitting comfortably using a disposable mouthpiece and nasal clip, with values of forced vital capacity (FVC), forced expiratory volume in the first second (FEV1), forced expiratory flow 25% -75% (FEF 25% -75%) and the FEV1 / FVC ratio. To perform the tests a portable spirometer (Micro Medical, Microloop, MK8, England) will be used and the values obtained will be interpreted according to the predicted values of Pereira el. al.
  These variables are being presented together because it is an examination called spirometry.
Respiratory Muscle Strength | 2 days
  The manovacuometry will be performed according to the recommendations of the American Thoracic Society and the European Respiratory Society (ATS / ERS) and the Brazilian Society of Pulmonology and Physiology (SBPC).
  The manovacuometry will be performed according to the recommendations of the American Thoracic Society and the European Respiratory Society (ATS / ERS) and the Brazilian Society of Pulmonology and Physiology (SBPC). Therefore, during the collection of MIP and MEP values, with the arms free and will be oriented to attach to your mouth a nozzle (type diver) with presence of leakage hole of 2mm of internal diameter.
  The individual will be instructed to perform a maximum expiration and maximal inspiration for at least 1,5s, so that the maximum sustained pressure for one second is observed (maximum mean pressure) in the manovacuometer MVD 300, Globalmed, Brazil.

CONTACTS AND LOCATIONS:
Locations (1):
- Daniella Cunha, Recife, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] WHO Expert Consultation. Appropriate body-mass index for Asian populations and its implications for policy and intervention strategies. Lancet. 2004 Jan 10;363(9403):157-63. doi: 10.1016/S0140-6736(03)15268-3. PMID 14726171
- [Result] Meier T, Luepschen H, Karsten J, Leibecke T, Grossherr M, Gehring H, Leonhardt S. Assessment of regional lung recruitment and derecruitment during a PEEP trial based on electrical impedance tomography. Intensive Care Med. 2008 Mar;34(3):543-50. doi: 10.1007/s00134-007-0786-9. Epub 2007 Jul 25. PMID 17653529
- See also: Related Info — http://pubmed.gov